CLINICAL TRIAL: NCT07241910
Title: A Phase I, Single-Center, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SYH2061 in Healthy Subjects
Brief Title: A Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SYH2061
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYH2061-001
Record Dates: First submitted 2025-11-17; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYH2061 group (Experimental): Subjects in experimental group will receive a single subcutaneous injection of SYH2061 on Day 1.
  Interventions: Drug: SYH2061
- Placebo group (Placebo Comparator): Subjects in placebo group will receive a single subcutaneous injection of placebo on Day 1.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYH2061 — subcutaneous injection
  Arms: SYH2061 group
Drug: Placebo — subcutaneous injection
  Arms: Placebo group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single-ascending dose study in healthy subjects to evaluate the safety, tolerability, PK, and PD of SYH2061.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be informed of the study before it begins, fully understand the study content, procedures, and potential adverse reactions, and voluntarily sign the written ICF;
2. Healthy male or female subjects, aged 18 to 55 years (inclusive);
3. Body mass index ranging from 19.0 to 28.0 kg/m2 (inclusive), with a body weight of ≥ 50 kg for males and ≥ 45 kg for females;
4. The results of various examinations, such as physical examination, vital signs, ECG, chest X-ray, abdominal B-scan ultrasound, and laboratory tests at screening are normal or abnormal without clinical significance;
5. Vaccinated against meningococcal ACYW135 vaccine and pneumococcal vaccine at least 14 days prior to the first dose, or have valid documentation of receiving the respective vaccinations within the past 3 years prior to dosing as evaluated by the investigator.;
6. Subjects and their partners agree to use effective and reliable contraceptive methods from 14 days before signing the ICF until 6 months after drug administration; male subjects agree not to donate sperm and female subjects agree not to donate ova from signing the ICF until 6 months after study drug administration;
7. Subjects are able to communicate well with the investigator and can complete the study in accordance with the protocol.

Exclusion Criteria:

1. History and/or current presence of clinically significant medical conditions, including but not limited to circulatory system disorders, hematological or hematopoietic system disorders, respiratory disorders, endocrine disorders, urinary system disorders, digestive system disorders, neurological or psychiatric disorders, autoimmune diseases, malignant tumors, severe trauma, or any other disease that should be excluded or may interfere with the interpretation of the study results in the opinion of the investigator;
2. History of splenectomy, or functional or anatomical asplenia;
3. Known or suspected hereditary or acquired complement deficiency or impaired complement activity, or complement activity below the normal range at screening;
4. History of meningococcal infection, or positive Neisseria meningitides test at screening;
5. Subjects who are frequently exposed to Neisseria meningitides (e.g., research, industrial, or clinical laboratory personnel, military personnel during recruit training, daycare center staff, etc.), and those who have traveled to or plan to travel to endemic areas for meningococcal meningitis (e.g., India, sub-Saharan Africa, Saudi Arabia) within 6 months before dosing or during the course of the study;
6. History of recurrent or chronic infections (e.g., recurrent upper respiratory tract infection, diarrhoea, etc.) or infections requiring systemic antibiotic therapy within 3 months before dosing;
7. Presence or suspicion of active viral, bacterial, fungal, or parasitic infection including herpes, herpes zoster, or cold sores within 14 days before dosing;
8. History or current presence of latent or active pulmonary tuberculosis, or positive T-SPOT test at screening;
9. History of major surgery within 6 months prior to screening, or plan to undergo major surgery during the course of the study;
10. Subjects with severe allergic diseases or allergic constitution (≥ 3 drug or food allergies), or a known history of allergy to the investigational drug components, oligonucleotide drugs, or vaccinations;
11. Subjects who are allergic to β-lactam antibiotics (e.g., penicillin, cephalosporins) or ciprofloxacin, or have any contraindications, or unwilling to use antibiotic prophylaxis as specified in the protocol;
12. Intolerance to subcutaneous injection, or presence of abdominal scars (from surgery, burns, etc.) that affect subcutaneous administration, and any skin abnormalities and/or tattoos that may affect the safety assessment of the injection site;
13. Any of the following liver function test results: alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin (TBIL), γ-glutamyl transferase (GGT), or alkaline phosphatase (ALP) above the upper limit of normal at screening;
14. Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m2 (calculated by the simplified MDRD formula) at screening;
15. Prolonged QT/QTc interval at screening or baseline (QTcF > 450 ms for males, > 470 ms for females);
16. Positive result for any of the following: hepatitis B surface antigen (HBsAg), hepatitis C virus antibody, human immunodeficiency virus (HIV) antigen/antibody, or Treponema pallidum antibody;
17. Use of any prescription drugs, over-the-counter drugs, herbal medicines or vitamin and dietary supplements within 14 days or 5 half-lives (whichever is longer) before dosing;
18. Received complement inhibitor treatment (e.g., Eculizumab, Crovalimab, etc.) within 6 months or 5 half-lives (whichever is longer) before dosing;
19. Received live or live-attenuated vaccines within 28 days before dosing, or plan to receive such vaccines during the course of the study (except for vaccinations planned by the study protocol);
20. Blood loss or blood donation of more than 200 mL within 3 months before screening (except for menstruation in females), or platelet donation within 2 weeks before screening;
21. History of drug abuse, or use of illicit drugs within 3 months before screening, or habitual use of any psychotropic drugs (including herbal medicines), or a positive urine drug screen;
22. Regular alcohol consumption within 6 months before screening, defined as weekly alcohol consumption exceeding 14 units (1 unit = 360 mL of 5% alcohol beer or 45 mL of 40% alcohol spirits or 150 mL of 12% alcohol wine), or inability to stop alcohol intake as required by the protocol during the study, or a positive blood alcohol test;
23. Average daily smoking of more than 5 cigarettes (or an equivalent amount of tobacco in e-cigarettes) within 3 months before screening, or unwilling to avoid using any tobacco products as required by the protocol during the study;
24. Participation in any clinical trial within 3 months before screening (or within 12 months before screening for oligonucleotide drugs)
25. In addition to the above requirements, female subjects who meet the following criteria should also be excluded: a. Pregnant or lactating women; b. Use of oral contraception within 28 days prior to screening; c. Use of long-acting estrogen and/or progesterone injections and/or implants within 6 months prior to screening; d. females of childbearing potential who had unprotected sexual intercourse with their partner within 28 days prior to dosing.
26. Any other conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2026-11-24 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with Adverse Events as Assessed by CTCAE v5.0 | Up to Day 337
  To assess the safety and tolerability of SYH2061 in healthy subjects

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of SYH2061 | Up to 72 hours post-dose
  To characterize the Cmax of SYH2061 in healthy subjects
Time to maximum observed plasma concentration (Tmax) of SYH2061 | Up to 72 hours post-dose
  To characterize the Tmax of SYH2061 in healthy subjects
Area under the concentration-curve from zero to the last quantifiable concentration (AUClast) of SYH2061 | Up to 72 hours post-dose
  To characterize the AUClast of SYH2061 in healthy subjects
Area under the concentration-time curve from zero to infinity (AUCinf) of SYH2061 | Up to 72 hours post-dose
  To characterize the AUCinf of SYH2061 in healthy subjects
Terminal elimination half-life (t1/2) of SYH2061 | Up to 72 hours post-dose
  To characterize the t1/2 of SYH2061 in healthy subjects
Apparent clearance (CL/F) of SYH2061 | Up to 72 hours post-dose
  To characterize the CL/F of SYH2061 in healthy subjects
Apparent volume of distribution (Vz/F) of SYH2061 | Up to 72 hours post-dose
  To characterize the Vz/F of SYH2061 in healthy subjects
Percent change from baseline in complement C5 and its fragments C5a and C5b-9 | Up to Day 337
  To assess the PD effects of SYH2061 in healthy subjects
Percent change from baseline in complement alternative pathway (CAP) | Up to Day 337
  To assess the PD effects of SYH2061 in healthy subjects
Percent change from baseline in complement classical pathway (CCP) | Up to Day 337
  To assess the PD effects of SYH2061 in healthy subjects
Incidence of ADA | Day85
  To assess the immunogenicity of SYH2061 in healthy subjects